CLINICAL TRIAL: NCT03037346
Title: Preparing Patients and Family Caregivers for Medical Decision Making: Evaluating the Impact of a Systematic Social Work Driven Approach on Medical Power of Attorney Documentation, Knowledge, Attitudes and Beliefs
Brief Title: Impact of a Systematic Social Work Driven Approach on Medical Power of Attorney Documentation, Knowledge, Attitudes, and Beliefs in Participants With Stage I-IV Gynecological Cancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2016-0704; NCI-2018-01745 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2016-0704 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-01-27; First posted 2017-01-31 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Caregiver; Malignant Female Reproductive System Neoplasm
MeSH Terms: interventions — Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Supportive Care (questionnaires, educational video) (Experimental): Participants (patients and family caregiver/MPOA) complete questionnaires about knowledge, attitudes, and beliefs of MPOAD. Participants without a MPOAD watch a 4-minute educational video about the importance of the role of MPOA.
  Interventions: Other: Questionnaire Administration; Other: Video

INTERVENTIONS:
Other: Questionnaire Administration — Complete questionnaires about MPOAD
Other: Questionnaire Administration — Ancillary studies
Other: Video — Watch educational video

SUMMARY:
This trial evaluates the impact of a systemic social work driven approach on medical power of attorney documentation, knowledge, attitudes, and beliefs in participants with stage I-IV gynecological cancers. Social work counseling and education may help increase the number of participants who complete medical power of attorney documents. Counseling and education may also affect attitudes about decision-making and willingness to take part in these conversations in participants with stage I-IV gynecological cancers and their family members and/or caregivers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate medical power of attorney documents (MPOAD) completion rate after a systematic social work counseling and education clinical process.

SECONDARY OBJECTIVES:

I. To determine change in medical power of attorney (MPOA)/primary family caregivers' knowledge, attitudes and beliefs about conditions for quality surrogate medical decision-making (MDM).

II. To determine change in MPOA/primary family caregivers' knowledge of patients' values and goals for MDM.

III. Evaluate patients' and MPOA/primary family caregivers' willingness to participate in future advance care planning discussions to discuss patients' values and goals important to MDM.

IV. Evaluate predictors of patient subgroups most likely to respond to the social work counseling and education clinical process.

V. Explore aspects of the Spanish language version of the advance care planning engagement survey to inform future validation studies.

OUTLINE:

Participants (patients and family caregiver/MPOA) complete questionnaires about knowledge, attitudes, and beliefs of MPOAD. Participants without a MPOAD watch a 4-minute educational video about the importance of the role of MPOA.

After completion of intervention, participants are followed up at 3 months.

ELIGIBILITY:
Inclusion Criteria:

* PATIENTS
* Diagnosis of invasive gynecologic malignancy stages 1-4.
* New patient in the Gynecologic Oncology Center.
* Adequate capacity to understand and complete MPOAD in the opinion of the study investigator or research assistant.
* Able to speak and understand English and/or Spanish.
* Provision of Institutional Review Board (IRB)-approved informed consent.
* Available MPOA or primary family caregiver who consents to study participation.
* FAMILY CAREGIVER/MPOA
* MPOA or if none documented in electronic health record (EHR), primary family caregiver, as designated by the patient.
* Permission to contact provided by patient.
* Adequate capacity to understand and complete study measures in the opinion of the study investigator or research assistant.
* Provision of IRB-approved informed consent.

Exclusion Criteria:

* Without a MPOA or available family caregiver.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 731 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2024-12-16 (Actual); Study Completion 2024-12-16 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who decline to participate in the study | Up to 3 months
  Will be reported with 95% confidence intervals. Descriptive demographic and disease characteristics for patients who decline study participation but allow collection of demographic and disease characteristics will be compared to those of participating patients.
Proportion of patients who already have medical power of attorney (MPOAD) at consult | Up to 3 months
  Will be reported with 95% confidence intervals. Baseline and changes in MPOA/primary family caregivers' knowledge, attitudes and beliefs about conditions for quality surrogate medical decision-making (MDM), in patients/primary family caregivers' self-efficacy and readiness for MPOA, and in patients/Primary family caregivers' knowledge of patients' values and goals for MDM, will be summarized and compared among the four patient groups: 1) had MPOAD at the consult already, 2) complete MPOAD at the first visit, 3) complete MPOAD after initial social work counselor visit and by 3 months, 4) do not complete MPOAD by 3 months, using Kruskal-Wallis test for continuous variables and either Chi-square test or Fisher's exact test for discrete variables, whenever appropriate. Univariate/multi-covariate logistic regression will be employed to evaluate the effect of potential factors on completion of MPOAD.
Proportion of patients who completed MPOAD at the first social work counselor visit | Up to 3 months
  Will be reported with 95% confidence intervals. Baseline and changes in MPOA/primary family caregivers' knowledge, attitudes and beliefs about conditions for quality surrogate MDM, in patients/primary family caregivers' self-efficacy and readiness for MPOA, and in patients/Primary family caregivers' knowledge of patients' values and goals for MDM, will be summarized and compared among the four patient groups: 1) had MPOAD at the consult already, 2) complete MPOAD at the first visit, 3) complete MPOAD after initial social work counselor visit and by 3 months, 4) do not complete MPOAD by 3 months, using Kruskal-Wallis test for continuous variables and either Chi-square test or Fisher's exact test for discrete variables, whenever appropriate. Univariate/multi-covariate logistic regression will be employed to evaluate the effect of potential factors on completion of MPOAD.
Proportion of participants who completed MPOAD after the first educational video | Up to 3 months
  Will be reported with 95% confidence intervals. Baseline and changes in MPOA/primary family caregivers' knowledge, attitudes and beliefs about conditions for quality surrogate MDM, in patients/primary family caregivers' self-efficacy and readiness for MPOA, and in patients/Primary family caregivers' knowledge of patients' values and goals for MDM, will be summarized and compared among the four patient groups: 1) had MPOAD at the consult already, 2) complete MPOAD at the first visit, 3) complete MPOAD after initial social work counselor visit and by 3 months, 4) do not complete MPOAD by 3 months, using Kruskal-Wallis test for continuous variables and either Chi-square test or Fisher's exact test for discrete variables, whenever appropriate. Univariate/multi-covariate logistic regression will be employed to evaluate the effect of potential factors on completion of MPOAD.
Proportion of participants who completed MPOAD within 3 months after the educational video | Up to 3 months
  Will be reported with 95% confidence intervals. Baseline and changes in MPOA/primary family caregivers' knowledge, attitudes and beliefs about conditions for quality surrogate MDM, in patients/primary family caregivers' self-efficacy and readiness for MPOA, and in patients/Primary family caregivers' knowledge of patients' values and goals for MDM, will be summarized and compared among the four patient groups: 1) had MPOAD at the consult already, 2) complete MPOAD at the first visit, 3) complete MPOAD after initial social work counselor visit and by 3 months, 4) do not complete MPOAD by 3 months, using Kruskal-Wallis test for continuous variables and either Chi-square test or Fisher's exact test for discrete variables, whenever appropriate. Univariate/multi-covariate logistic regression will be employed to evaluate the effect of potential factors on completion of MPOAD.
Willingness to participate in future advance care planning discussions | Up to 3 months
  Willingness to participate in future Advance Care Planning discussions for patients' values and goals important to MDM will be tabulated.

CONTACTS AND LOCATIONS:
Overall Officials: Donna S Zhukovsky, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org